CLINICAL TRIAL: NCT05911685
Title: A Prospective, Multicenter, Single-arm Objective Performance Criteria Evaluation of the Safety and Efficacy of a Novel SeaLA™ Left Atrial Appendage Occluder in Patients With Nonvalvular Paroxysmal Atrial Fibrillation
Brief Title: Evaluation of the Safety and Efficacy of a Novel SeaLA™ Left Atrial Appendage Occluder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hangzhou Dinova EP Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAA01
Record Dates: First submitted 2023-06-06; First posted 2023-06-22 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Left atrial appendage occlusion (Experimental)
  Interventions: Device: SeaLA™ left atrial appendage occluder

INTERVENTIONS:
Device: SeaLA™ left atrial appendage occluder — 1. Guided by esophageal ultrasound (TEE) and angiography, the diameter of the left atrial appendage anchoring zone and the longest depth of the left atrial appendage were measured to determine the appropriate size of the left atrial appendage occluder.
  2. Maintain Activated Clotting Time (ACT) greater than 250 seconds after atrial septal puncture to the completion of the entire procedure.
  3. Before the plugging device is released, confirm whether there is a residual peri-device leak, and if there is a residual peri-device leak, consider retracting the occluder to reposition the release or retract the occluder to choose a larger size occluder to re-occlusion. If ultrasound confirms residual peri-device leak greater than 5 mm, do not release and implant the left atrial appendage occluder.
  4. Before and after release, confirm the position and stability of the occluder under ultrasound (TEE), and confirm that the occluder completely occludes the left atrial appendage.

SUMMARY:
This study adapted a prospective, multicenter single-group objective performance criteria design. A total of 163 patients with non-valvular atrial fibrillation were enrolled in the clinical trial，follow up were scheduled in 7 days, 45 days, 6 months, 12 months, 2 years, 3 years, 4 years and 5years after procedure.

DETAILED DESCRIPTION:
This study adapted a prospective, multicenter single-group objective performance criteria design。A total of 163 patients with non-valvular atrial fibrillation were enrolled in the clinical trial, the patients signed the informed consent form and met the inclusion and exclusion criteria, the subjects were implanted with the SeaLA™ LAA (left atrial appendage) occlusion, and TTE(transthoracic echocardiography) examination was performed 7 days after procedure or before discharge (whichever comes first), TEE(transesophageal echocardiography) examination were performed 45 days and 6 months after procedure, and TTE examination at 12 months. In the 2nd, 3rd, 4th, and 5th years of telephone follow-up subjects, the main adverse event data were collected and analyzed, and the long-term safety and efficacy of the left atrial appendage closure device product after implantation were evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with nonvalvular paroxysmal, persistent or permanent atrial fibrillation;
2. Subject is not suitable for long-term treatment with anticoagulant;
3. CHA2DS2-VASC score（Atrial fibrillation stroke risk score） ≥ 2;
4. Subjects are suitable for dual antiplatelet therapy for 3 months and complete follow-up;

Exclusion Criteria:

1. Patients with atrial fibrillation caused by rheumatic heart valve disease, degenerative heart valve disease, or congenital heart valve disease;
2. Patients after heart transplantation;
3. Unstable angina or recent myocardial infarction < 3 months;
4. Cardiac function IV (NYHA grade);
5. Subject requires atrial fibrillation catheter ablation surgery within 30 days of LAA occlusion device implantation;
6. Excludes the case of atrial fibrillation catheter ablation and LAA closure in the same surgery (if atrial fibrillation catheter ablation and LAA closure are operated on the same operation, it is recommended to have catheter ablation before closure);
7. Subject has an electrical cardioversion plan within 30 days of LAA occlusion device implantation;
8. After mechanical prosthetic valve implantation;
9. History of stroke or TIA(transient ischemic attack) within 30 days;
10. Thrombocytopenia (platelets≤ 100.000 pcs/mcL);
11. Active endocarditis, sepsis;
12. Heart tumor or other malignant tumor, life expectancy < 1 year;
13. subjects who are pregnant, lactating or planning to become pregnant during clinical trials (must undergo a pregnancy test before surgery, except for women of non-childbearing age);
14. are currently participating in clinical trials of other drugs or medical devices and have not completed the primary endpoint of the study, which may cause confusion in the results of this study or may affect subjects' compliance with this study follow-up;
15. The subject is subordinate to the sponsor or clinical trial institution or investigator;
16. The investigator judged that the subject's compliance was poor and could not complete the clinical trial requirements;
17. Allergy to nitinol or contrast media;
18. There is a complex movable/ruptured/> 4mm atherosclerotic plaque at the ascending aorta/aortic arch;
19. Patients with symptomatic carotid artery stenosis (such as carotid artery stenosis greater than 50%);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2025-01-21 (Estimated)

PRIMARY OUTCOMES:
Left atrial appendage closure rate | 6 months after procedure
  After the closure device is implanted, it is confirmed by ultrasound that no forward or reverse blood flow passes through the closure device, and the residual forward or reverse blood flow at the edge of the closure device is ≤ 3mm

SECONDARY OUTCOMES:
Device success rate | immediately after the procedure
  smooth delivery of left atrial appendage occluder to left atrial appendage, successful release of left atrial appendage occlusion, smooth withdrawal of delivery system
Ischemic stroke rate | 12 months after the procedure
  Ischemic stroke refers to the loss of nerve function caused by transient ischemic attack, cerebral thrombosis or cerebral embolism caused by the brain itself and/or systemic blood circulation disorders leading to cerebral blood supply disorders. Ischemic stroke is defined as a modified Rankin score (mRS) ≥2 90 days after stroke onset. The scale runs from 0 to 5, running from perfect health without symptoms to death, higher scores mean a worse outcome, 0 means no symptoms, 5 means dead.
Major adverse events rate | 7 days after procedure
  Unexplained death or any device- or procedure-related complications, including but not limited to: death, severe cardiac tamponade requiring pericardiocentesis or surgery, instrument embolism, surgery-related stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of the Northern Theater of the Chinese People's Liberation Army, Shengyang, China

REFERENCES:
- [Derived] Wang Z, Chu H, Chen X, Tao L, Yuan Y, Ru L, Wang J, Fan Y, Hu H, Wang C, Chen M, Huang W, Zhou D, Liu X, Liang M, Liu J, Han Y. Percutaneous left atrial appendage closure with SeaLA device in non-valvular atrial fibrillation. Catheter Cardiovasc Interv. 2024 Dec;104(7):1491-1498. doi: 10.1002/ccd.31056. Epub 2024 Jun 6. PMID 38841867